CLINICAL TRIAL: NCT00853281
Title: A Cluster Randomized Trial to Evaluate the Effectiveness of Long Lasting Insecticidal Hammocks for Controlling Forest Malaria in Central Vietnam
Brief Title: A Cluster Randomized Trial to Evaluate Long Lasting Insecticidal Hammocks to Prevent Forest Malaria in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: National Institute of Malariology, Parasitology and Entomology, Vietnam (Other Government); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Umberto D'Alessandro, MD, Institute of Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LLIH
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Malaria
Keywords: Forest malaria prevention; Long-lasting insecticidal hammocks; Cluster randomized trial; Central Vietnam
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hammocks with LLIN (Experimental): Locally-made hammocks covered with long-lasting insecticidal net (LLIN)- Olyset(R), used in addition to the standard vector control measures
  Interventions: Other: Hammocks with LLIN
- ITN (Active Comparator): Standard vector control measures (insectice-treated net or ITN)
  Interventions: Other: Standard vector control measures

INTERVENTIONS:
Other: Hammocks with LLIN — Locally-made hammocks covered with long lasting insecticidal nel (LLIN)
  Other Names: Oliset(R)
  Arms: Hammocks with LLIN
Other: Standard vector control measures — Insectice-treated net
  Other Names: ITN
  Arms: ITN

SUMMARY:
In Central Vietnam, forest malaria remains difficult to control due to the complex interactions between human, vector and environmental factors. Untreated bednets had a significantly protecting effect for villagers, except for those regularly sleeping in the forest, who suffer a significantly higher number of clinical attacks. Thus, there is need to target this high-risk group with new intervention based on long-lasting insecticidal materials. Hammocks are extensively used by people working in the forest, therefore long-lasting insecticidal hammocks (LLIH) could achieve a good individual protection.

The Investigators proposed to evaluate their effectiveness in a community-based trial, comparing them to the standard vector control methods (insecticide-treated nets).

DETAILED DESCRIPTION:
In Central Vietnam, forest malaria remains difficult to control due to the complex interactions between human, vector and environmental factors. A community-based study carried out between 1999 and 2001 showed that regular forest activity was a strong risk factor for malaria infection. Untreated bednets had a significantly protecting effect for villagers, except for those regularly sleeping in the forest, who suffered a significantly higher number of clinical attacks. Thus, there is need to target this high-risk group with new intervention based on long-lasting insecticidal materials. Hammocks are extensively used by people working in the forest, therefore long-lasting insecticidal hammocks (LLIH) could achieve a good individual protection.

The Investigators proposed to evaluate their effectiveness in a community-based trial, comparing them to the standard vector control methods (insecticide-treated nets): communities have been grouped into clusters of about 1000 înhabitants, and clusters were randomized to either the active intervention or the active control, and followed up for 24 month.

ELIGIBILITY:
Inclusion Criteria:

* All residents in the 20 concerned study clusters and willing to give informed consent to participate

Exclusion Criteria:

* People not willing to give informed consent to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18646 (Actual)
Dates: Start 2004-03; Primary Completion 2006-12 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Reduction of malaria prevalence and incidence | 24 months

SECONDARY OUTCOMES:
Reduction of malaria sero-prevalence | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Annette Erhart, MD, Study Director — Institute of Tropical Medicine
Locations (1):
- Ninh Thuan Provincial Malaria Station, Phan Rang-Tháp Chàm, Ninh Thuan, Vietnam

REFERENCES:
- [Derived] Thang ND, Erhart A, Speybroeck N, Xa NX, Thanh NN, Ky PV, Hung le X, Thuan le K, Coosemans M, D'Alessandro U. Long-Lasting Insecticidal Hammocks for controlling forest malaria: a community-based trial in a rural area of central Vietnam. PLoS One. 2009 Oct 7;4(10):e7369. doi: 10.1371/journal.pone.0007369. PMID 19809502